CLINICAL TRIAL: NCT04729816
Title: Assessing the Dose Response of a Lead Fiber Snack Prototype on the Gut Microbiome and Host Metabolome and Proteome
Brief Title: Assessing the Dose Response of a Lead Fiber Snack Prototype
Acronym: FDR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 202010046
Record Dates: First submitted 2020-11-09; First posted 2021-01-29 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Microbiota; Gastrointestinal Microbiome
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Fiber supplementation increasing by 10.2g per 2-week dosing period, from 0 to 30.6g supplemental fiber at the end of the dose escalation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary Intervention (Experimental): All participants will stay weight stable while undergoing 5 phases of a dietary intervention that lasts 62 days.
  Interventions: Other: Controlled, high fat/low fiber diet background diet, sequentially supplemented with an escalating dose of a fiber-blend snack food.

INTERVENTIONS:
Other: Controlled, high fat/low fiber diet background diet, sequentially supplemented with an escalating dose of a fiber-blend snack food. — Phase 1: Participants will be provided with a high fat/low fiber diet in the form of packed out meals and snacks for 10 days in total (days 2-11 and days 54-63)
  Phase 2: Participants will be provided with the high fat/low fiber diet, plus 1 daily fiber-blend snack serving from days 12-25
  Phase 3: Participants will receive 2 daily fiber-blend snack servings to supplement the high fat/low-fiber diet from days 26-39.
  Phase 4: Participants will receive 3 daily fiber-blend snack servings to supplement the high fat/low-fiber diet from days 40-53.
  Phase 5: Participants will return to the unsupplemented high fat/low fiber diet for days 54-63

SUMMARY:
Aim: To test the effects of a fiber-blend containing snack prototype in an escalating dose regimen (from 1 to 3 servings per day over a period of 6 weeks) on the configuration and gene content of the gut microbiota of overweight and obese participants (BMI 25-35 kg/m2), while consuming a controlled diet that contains quantities of saturated fats in the upper tertile and quantities of fruits and vegetables in the lower tertile of consumption in the NHANES database (high saturated fat-low fruit and vegetable; HiSF-LoFV). Changes in the representation of bacterial genes involved in carbohydrate utilization in the microbiomes of participants will be correlated with changes in plasma biomarkers at the end of each escalating dose phase by comparing features of their pre- vs post-treatment plasma proteomes and metabolomes.

Design: Participants will be asked to continue to consume their habitual diet (free diet phase) for 1 day prior to being provided with a HiSF-LoFV diet in the form of packed-out meals and snacks to consume for the following 62 days. Ten days after starting to consume the HiSF-LoFV diet, participants will supplement this diet with a fiber-blend containing snack (~10g fiber/serving) once daily for a total of 14 days; the energy contribution from the HiSF-LoFV diet will be reduced accordingly to maintain energy needs during this time and the remainder of the study. For the next 14 days, the diet will be supplemented with two of the same fiber-blend containing snacks per day, followed by 14 days in which the snacks will be consumed three times daily. Subsequently, a 'wash-out' phase of ten days in which the HiSF-LoFV diet is consumed without any of fiber snack supplementation will conclude the study. Stool, urine and blood will be sampled periodically throughout.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥25.0 and ≤35.0 kg/m2

Exclusion Criteria:

* Previous bariatric surgery
* Significant organ system dysfunction (e.g. diabetes, severe pulmonary, kidney, liver, or -cardiovascular disease)
* Cancer or cancer that has been in remission for less than 5 years
* Major psychiatric illness
* Inflammatory gastrointestinal disease
* Pregnant or lactating women
* Use of medications that are known to affect the study outcome measures
* Use of medications or supplements known to affect composition of the gut microbiota within the last 30 days (e.g. antibiotics)
* Bowel movements less than 3 times per week
* Vegans, vegetarians, and those with allergies, aversions, or sensitivities to foods provided in the study
* Persons that are not able to grant voluntary informed consent
* Persons who are unable or unwilling to follow the study protocol or who the research team deems not an appropriate candidate for the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Changes to the gut microbiota/microbiome | Stool samples will be collected periodically from day 1 through the final day of the 63-day study
  Changes to the gut microbiota/microbiome as a function of background diet and fiber dose escalation using culture independent methods. Investigators will use higher order singular value decomposition (HOSVD) to analyze changes in the gut microbiome - including the representation of carbohydrate-active enzyme genes (CAZymes), metabolic pathways and Amplicon Sequence Variants (ASVs) in shotgun sequencing datasets generated from fecal DNA collected at the beginning and end of each dose escalation phase.
Changes in the plasma proteome/metabolome | Fasted blood draws will be collected at day 1, day 11, day 25, day 39, day 53, and day 63. Stool samples will be collected periodically from day 1 through the final day of the 63-day study
  Changes in the plasma proteome/metabolome (aptamer-based proteomics/mass spectrometry) as a function of fiber dose escalation and their correlation with features of the gut microbiome using cross-correlation singular value decomposition (CC-SVD).
Change in plasma lipid profile | Fasted blood draws will be collected at screening, day 11, day 25, day 39, day 53, and day 63
  Changes in the plasma lipid profile as a function of background diet and fiber dose escalation as assessed by complete metabolic and lipid panels.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Patnode ML, Beller ZW, Han ND, Cheng J, Peters SL, Terrapon N, Henrissat B, Le Gall S, Saulnier L, Hayashi DK, Meynier A, Vinoy S, Giannone RJ, Hettich RL, Gordon JI. Interspecies Competition Impacts Targeted Manipulation of Human Gut Bacteria by Fiber-Derived Glycans. Cell. 2019 Sep 19;179(1):59-73.e13. doi: 10.1016/j.cell.2019.08.011. PMID 31539500